CLINICAL TRIAL: NCT02258698
Title: Insulin Sensitivity, Irisin and Adipokines as Outcome Parameters in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: McGill University (Other)
Responsible Party: Sponsor
Other Study IDs: 56/13
Record Dates: First submitted 2014-09-29; First posted 2014-10-07 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Insulin Resistance; Diabetes Mellitus Type 2; Other Functional Disturbances Following Cardiac Surgery
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (Serum)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elective on-pump cardiac surgery: Observation of perioperative Insulin resistance in patients undergoing elective on-pump cardiac surgery (CABG and/or valve repair)
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Blood samples for assessing Insulin resistance by HOMA, QUICKI, HbA1c, ANGPTL2, CXCL5, visfatin and irisin are drawn during induction of anesthesia, upon arrival on the intensive care unit and on postoperative day 1 and 3. Thirty days after surgery adverse outcomes covering all-cause morbidity and mortality will be assessed.

SUMMARY:
BACKGROUND: Surgical injury and inflammation provoke a stereotypical stress response. Insulin resistance plays an intriguing role in these metabolic alterations and depends on the intensity of injury. Metabolic derangements resulting from peripheral insulin resistance are unambiguously related to adverse outcomes and higher perioperative complication rates. Therefore, insulin resistance offers to act as a marker for stress and is potentially relevant in predicting clinical outcome. Plasma-glycosylated hemoglobin A (HbA1c) is an established indicator for blood glucose control and has a prognostic value regarding outcomes after major surgical interventions.

Adipose tissue holds a key function in endocrine metabolism by releasing multiple substances, so-called adipose-derived secreted factors or adipokines. Recent studies have linked several adipokines to overall insulin sensitivity in metabolic syndrome-related conditions as well as in critical illness. Irisin, a recently identified myokine acts on white adipose tissue and plays a role in the prevention of insulin resistance.

AIMS OF THE STUDY: The aim of this study is to assess the level and the effects of perioperative insulin resistance on clinical outcome in cardiac surgery patients. Based on previous studies suggesting glucose homeostasis and insulin resistance are associated with severity of illness and outcome in critically ill patients,it is proposed that patients with marked insulin resistance suffer from worse clinical outcome. This study protocol evaluates the ability of homeostasis model assessment (HOMA), quantitative insulin sensitivity check index (QUICKI), HbA1c, the adipokines Angiopoietin-like protein 2 (ANGPTL2), C-X-C motif chemokine 5 (CXCL5), and visfatin, and the myokine irisin to indicate perioperative insulin resistance and explores for correlation with adverse clinical outcomes after 30 days.

MATERIAL & METHODS: 325 patients admitted to the surgical intensive care unit after elective on-pump cardiac surgery will be consecutively enrolled. Baseline characteristics and routine blood samples will be assessed the day before surgery. Study blood samples will be drawn preoperatively in the induction bay of anesthesia to measure the insulin resistance indices HOMA and QUICKI, HbA1c, ANGPTL2, CXCL5, visfatin, and irisin. Blood glucose, irisin, adipokines, and routine biochemical tests will be assessed upon admission to the intensive care unit and on postoperative days 1 and 3. Adverse outcomes will be assessed 30 days after surgery. Sample size is set to ensure at least 80% power at a significance level of 0.05.

DETAILED DESCRIPTION:
see Information below

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* Admission to the surgical intensive care unit after elective cardiac surgery (aortocoronary bypass and/or valve repair)
* Being capable of understanding and signing the consent form

Exclusion Criteria:

* Blood glucose values requiring continuous insulin infusion preoperatively
* Ongoing selenium therapy
* Pregnancy
* Interventional valve repair
* Intraoperative hypothermic cardiac arrest
* Off-pump cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 325 patients admitted to the surgical intensive care unit after elective on-pump cardiac surgery (Table 1) will be consecutively enrolled. This study population has been chosen not only because of the clinically relevant stress response to cardiac surgery but also because of the opportunity to differentiate between the different impacts of the cardiovascular system and the metabolic state on insulin resistance.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse outcomes in relation to Insulin resistance measured as HOMA (homeostasis model assessment) | 30 days after surgery

SECONDARY OUTCOMES:
Number of adverse outcomes in relation to Insulin resistance measured as QUICKI | 30 days after surgery
Number of adverse outcomes in relation to Insulin resistance measured as HbA1c | 30 days after surgery
Number of adverse outcomes in relation to Insulin resistance measured as ANGPTL2 | 30 days after surgery
Number of adverse outcomes in relation to Insulin resistance measured as CXCL5 | 30 days after surgery
Number of adverse outcomes in relation to Insulin resistance measured as NAMPT | 30 days after surgery
Number of adverse outcomes in relation to Insulin resistance measured as irisin | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kopp Lugli, MD, MSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Andrea Kopp Lugli, Basel, Canton of Basel-City, Switzerland